CLINICAL TRIAL: NCT02568592
Title: Exercise Substrate Utilisation and Endurance Performance Following Short-term Manipulation of Dietary Fat Intake in Women
Brief Title: Exercise Substrate Utilisation and Endurance Performance Following Short-term Manipulation of Dietary Fat Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ERN_15-0012
Record Dates: First submitted 2015-05-13; First posted 2015-10-06 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Fat (Experimental): High Fat - Carbohydrate (20%), Fat (65%), Protein (15%)
  Interventions: Dietary Supplement: High Fat
- Normal (Experimental): Normal - Carbohydrate (50%), Fat (35%) and Protein (15%)
  Interventions: Dietary Supplement: Normal
- Normal + Extra Fat (Experimental): Normal + Extra Fat - Carbohydrate (50%), Fat (65%), Protein (15%). Carbohydrate and protein intake identical in absolute amounts to NORM (Normal), with an additional 30% extra energy coming from fat.
  Interventions: Dietary Supplement: Normal + Extra Fat

INTERVENTIONS:
Dietary Supplement: High Fat — High Fat - Carbohydrate (20%), Fat (65%), Protein (15%)
  Arms: High Fat
Dietary Supplement: Normal — Normal - Carbohydrate (50%), Fat (35%) and Protein (15%)
  Arms: Normal
Dietary Supplement: Normal + Extra Fat — Normal + Extra Fat - Carbohydrate (50%), Fat (65%), Protein (15%). Carbohydrate and protein intake identical in absolute amounts to NORMAL, with an additional 30% extra energy coming from fat.
  Arms: Normal + Extra Fat

SUMMARY:
The capacity to burn fat as fuel for exercise may have important implications for sporting performance, with dietary fat intake positively influencing this ability.

Endurance performance and the ability to burn fat will be measured in women runners following the consumption of 3 diets varying in the amount of fat and carbohydrate.

DETAILED DESCRIPTION:
Dietary fat intake positively influences the ability to burn fat during exercise in women but not men, whereas carbohydrate intake negatively influences fat oxidation in both sexes. The independent nature of dietary fat intake as a predictor of the ability to burn fat in women suggests that in conditions of adequate carbohydrate intake providing additional fat may increase fat oxidation in women whereas it does not in men. It is of interest to explore if indeed women are responsive (i.e., increase in fat oxidation) to short-term increases in dietary fat intake induced by overfeeding (adequate carbohydrate) or if as appears to be the case in men reduced carbohydrate intake as typically employed in high-fat, low carbohydrate dietary studies is also a prerequisite for enhancing fat oxidation in women, and whether this translates into a difference in exercise endurance performance.

ELIGIBILITY:
Inclusion Criteria:

* BMI >17.0 < 25 kg/m2
* Good General Health
* Accustomed to vigorous physical activity
* Run > 2 times per week
* V̇O2max >50ml/kg/min
* Weight Stable > last 6months
* Non Smoker
* Pre-menopausal, and either eumenorrheic and regularly menstruating, or using monophasic hormonal oral contraceptives for > 3 months.

Exclusion Criteria:

* Currently taking part in another scientific/clinical study
* Taking any prescription drug / supplement thought to influence metabolism
* Following unusual dietary practices (such as intermittent fasting or low carbohydrate diets)
* Pregnant
* Breast Feeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Rates of fat oxidation during exercise | 90 minutes of sub-maximal exercise
  Rates of fat oxidation to be measured via indirect calorimetry during 90 minutes of submaximal exercise

SECONDARY OUTCOMES:
5km running performance | Immediately following measurement of Primary Outcome measure
  Time to complete 5km on a treadmill
Change in plasma glucose concentration | 90 minutes sub-maximal exercise
  Area under the plasma concentration versus time curve (AUC) of glucose
Change in Free Fatty Acid concentration | 90 minutes sub-maximal exercise
  Area under the plasma concentration versus time curve (AUC) of Free Fatty Acid
Change in plasma glycerol concentration | 90 minutes sub-maximal exercise
  Area under the plasma concentration versus time curve (AUC) of glycerol

CONTACTS AND LOCATIONS:
Overall Officials: Gareth A Wallis, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No